CLINICAL TRIAL: NCT02798094
Title: Stress Sensitivity and Reward Responsivity: An Integration of Two Endophenotypes in Major Depression
Brief Title: Stress Sensitivity and Reward Responsivity in Depression
Acronym: CAN-BIND-04
Status: Completed | Type: Observational
Sponsor: Dr. Kate Harkness (Other)
Collaborators: University Health Network, Toronto (Other); University of Calgary (Other); Harvard University (Other); McGill University (Other)
Responsible Party: Sponsor-Investigator, Dr. Kate Harkness, Dr., Queen's University
Organization: Queen's University (Other)
Other Study IDs: PSYC-154-14
Record Dates: First submitted 2016-05-13; First posted 2016-06-14 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Depressed
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva is collected at eight points across the second session in 5mL vials. Saliva samples are assayed for neuroendocrine hormones (e.g., cortisol). Whole blood is collected in EDTA tubes at the first session. Whole blood is currently being banked. No assays are being conducted at this time.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Depressed Participants: No intervention
- Healthy Control Participants: No intervention

SUMMARY:
The goal of this project is to learn more about the different ways in which people process information that is stressful and rewarding, and how abnormalities in these two processes are related to depression.

DETAILED DESCRIPTION:
Participants will participate in two 3-hour sessions separated by a week at Providence Care, Mental Health Services, and a third, 1.5-hour session at the Queen's MRI Facility. At the first session participants will complete a packet of questionnaires about their mood and take part in an interview about their mood, medications, drug use, and any other symptoms, as well as an interview about their relationships with their parents and any experiences of abuse. At the second session participants will participate in a stress test, which involves giving a speech to a panel. The investigators will also collect saliva samples to look at stress hormones. Participants will also complete a task on the computer that involves looking at cartoon faces and making decisions about them. At the third session, the investigators take images of of participant's brain using a magnetic resonance scanner.

Participants are invited to participate in a 6-month follow-up for this study, which would involve the same procedure as outline above.

ELIGIBILITY:
For Depressed Participants:

Inclusion Criteria:

* Outpatients aged 18-65
* Currently suffering from unipolar depression
* Fluency in English, sufficient to complete the interviews and self-report questionnaires

Exclusion Criteria:

* Clinical diagnosis of bipolar disorder, psychotic disorders, current alcohol/substance dependence, or significant medical comorbidity
* Treatment-resistant (defined as failing more than 3 trials of anti-depressant medication)
* History of neurological insult (e.g., concussion), neurological disease, seizure disorder
* Smokers
* Pregnant women
* Endocrine disorders
* High suicidal risk, defined by clinician judgement

For Healthy Control Participants:

Inclusion Criteria:

* Adults aged 18-65
* No history of Axis I disorders according to DSM-IV-TR criteria, as determined by the SCID
* No first-degree relatives diagnosed with bipolar disorder
* Fluency in English, sufficient to complete the interviews and self-report questionnaires

Exclusion Criteria:

* History of neurological insult (e.g., concussion), neurological disease, seizure disorder
* Smokers
* Pregnant women
* Endocrine disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 219 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Stress Sensitivity: Salivary Hormone and Stress Challenge Test (TSST) | 2 hours after beginning of Time B Appointment
  Participants are required to give a speech and an arithmetic test in front of a panel. Saliva samples are collected at 8 points throughout the test.

SECONDARY OUTCOMES:
Mood and Anxiety Symptom Questionnaire (MASQ) | Administered at first baseline appointment and covers past 2 weeks
  Self-report scale of general distress (GD), anhedonic depression (AD), and anxious arousal (AA) symptoms
Reward Responsivity: Probabilistic Reward Task | Administered at second baseline appointment
  Computerized task that requires participants to choose between two stimuli and develop a response bias to the more frequently rewarded stimulus.
Snaith Hamilton Pleasure Scale (SHAPS and SHAPS-C) | Administered at first baseline appointment and covers past 2 weeks prior to interview
  Self-report of anhedonia symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Kate Harkness, PhD, Principal Investigator — Queens University
Locations (1):
- Queen's University, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided